CLINICAL TRIAL: NCT06606405
Title: Serratus Anterior Activation and Its Relationship with Shoulder Rotators in Adolescent Volleyball Players with Scapular Dyskinesia During Plank Exercise
Brief Title: The Activation of Serratus Anterior Muscle During the Plank Exercise
Status: Completed | Type: Observational
Sponsor: Berivan Beril Kılıç (Other)
Responsible Party: Sponsor-Investigator, Berivan Beril Kılıç, Asst. Prof., Biruni University
Organization: Biruni University (Other)
Other Study IDs: 69869
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Scapular Dyskinesis
Keywords: scapular dyskinesis; plank exercise; serratus anterior; shoulder rotator strength; athlete

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Scapular Dyskinesis Group: adolescent volleyball players with scapular dyskinesis
  Interventions: Diagnostic Test: scapular dyskinesis test
- Control Group: adolescent volleyball players without scapular dyskinesis
  Interventions: Diagnostic Test: scapular dyskinesis test

INTERVENTIONS:
Diagnostic Test: scapular dyskinesis test — Scapular dyskinesia in athletes will be visually evaluated. It will be considered present if, during 3 out of 5 arm elevation attempts, any of the following are observed: prominence of the medial or upper scapular border, lower scapular angle, excessive clavicular elevation, or rapid downward rotation of the scapula. After the tester demonstrates the required movements, the athletes will practice the movement. The test will begin with the arms at the sides of the body, elbows straight, and shoulders in neutral rotation. Two testers will observe from behind and video record the movements. Participants will be instructed to raise their arms as high as possible simultaneously, using the 'thumbs up' position, and to maintain this position for 3 seconds before lowering their arms for another 3 seconds. Athletes will perform the arm elevation with a dumbbell weight calculated as 1.4% of their body weight (Kamonseki, Haik, Ribeiro, Almeida, & Camargo, 2023).

SUMMARY:
Scapular dyskinesia is a condition characterized by changes in the resting position or movement of the scapula, which can impair shoulder function. Issues such as increased glenohumeral angle, reduced rotator cuff strength, and decreased subacromial space are commonly observed in athletes and sedentary individuals. Scapular muscle imbalances, particularly in the serratus anterior and lower trapezius muscles, are key contributors to dyskinesia. Studies show decreased EMG activity in these muscles among sedentary individuals, while increased activity is noted in overhead athletes. The relationship between serratus anterior activity and shoulder external rotation strength varies, highlighting the importance of strengthening scapular muscles to prevent injury in athletes.

The core, including the spine, hips, pelvis, and abdomen, provides stability and transfers forces throughout the body. Core and scapular stability are interrelated, and impairment in scapular stability can weaken core strength, increasing the risk of injury. Therefore, exercises targeting both the core and scapular muscles are vital in athletic training programs. The plank exercise, which minimizes spinal load and promotes strength, is preferred for enhancing both core and scapular endurance. However, improper form, especially due to weak stabilizer muscles, can lead to compensations that increase injury risk, such as long thoracic nerve injury. Although studies exist on serratus anterior activity during plank exercises, there is limited research on its activation in athletes with scapular dyskinesia.

DETAILED DESCRIPTION:
Scapular dyskinesia is defined as changes in the resting position of the scapula or in scapular movement. This condition can lead to negative changes in optimal shoulder function in individuals (Huang, Chen, Du, & Lin, 2020; Jildeh, Ference, Abbas, Jiang, & Okoroha, 2021). Changes such as an increase in the glenohumeral angle during horizontal abduction with scapular dyskinesia, a decrease in the maximal strength of the rotator cuff muscles responsible for compression stability, and a decrease in the subacromial space during overhead functions have been reported (Kibler & Sciascia, 2019). These resulting functional impairments and imbalances are observed in 67-100% of athletes, as well as sedentary individuals, sometimes without symptoms and sometimes accompanied by shoulder pathology (Silva et al., 2022). While many factors contributing to the development of scapular dyskinesia have been identified, one key factor is scapular muscle imbalances. The scapulothoracic muscle groups frequently emphasized in relation to scapular dyskinesia are the lower trapezius and serratus anterior. The serratus anterior muscle is responsible for upward rotation, external rotation, and posterior tilt of the scapula. This muscle is crucial for maintaining normal alignment and the continuity of functional scapular movement (Ludewig, Cook, & Nawoczenski, 1996; Ludewig & Reynolds, 2009). In a study conducted with sedentary individuals, it was reported that the EMG activity of the lower trapezius and serratus anterior muscles decreased in the presence of scapular dyskinesia (Ann MJ Cools et al., 2014). In contrast to this study, the EMG activity of the serratus anterior muscle in overhead athletes with scapular dyskinesia was examined during various movement patterns and functions such as shoulder elevation, push-up exercises, and tennis serves. It was suggested that muscle activity increased compared to sedentary individuals, and this increase should be further investigated in the future (de Paula Marques & Dionisio, 2024). Another point emphasized is the relationship between serratus anterior muscle activation and shoulder external rotation force in individuals with dyskinesia. While it has been stated that serratus anterior muscle activity decreases in the presence of scapular dyskinesia, external rotation muscle strength varies depending on the evaluated position. The importance of scapular muscles for shoulder external rotation strength has also been highlighted (Uga, Nakazawa, & Sakamoto, 2016). Strengthening the muscles responsible for external rotation in overhead athletes and restoring normal scapular movement are key points that should be emphasized as a whole in injury prevention programs (Ann M. Cools, Johansson, Borms, & Maenhout, 2015; Tooth et al., 2020).

The core region of the body includes the spine, hips, pelvis, proximal lower extremities, and abdomen (Kibler, Press, & Sciascia, 2006). The strength of these muscles allows for the transfer of compressive, translational, and shear forces, which serve to mechanically stabilize the spine and distribute forces to the rest of the body (Akuthota, Ferreiro, Moore, & Fredericson, 2008; Fredericson & Moore, 2005). Core stability is defined as the ability to control the position and movement of the trunk over the pelvis during integrated kinetic chain activities. It allows for the optimal transfer and control of force and movement to the terminal segment. Similar to the core muscles, the scapula plays an important role in transferring the force produced to the distal segments. Impairment in scapular stability can lead to a decrease in core strength, thereby increasing the risk of injury and reducing athletic performance. For this reason, exercises aimed at increasing scapular muscle and core endurance should be incorporated into athletes' exercise programs to prevent injury and enhance performance (Cobanoglu, Keklik, Zorlular, Polat, & Akaras, 2019). One of the exercises frequently included in Korean strength training programs for athletes is the plank exercise. Unlike sit-up exercises, the plank exercise is widely preferred to increase strength and endurance because it does not place a load on the lumbar spine and only minimally loads the spine when performed using body weight (Topçu et al., 2022). It is very important to perform plank exercises with correct segment alignment. The correct plank position is achieved in a push-up stance, with body weight supported by the forearms, elbows, and toes. The arms should be placed directly under the shoulder joints, and the entire body should maintain a straight alignment (Neporent, Schlosberg, & Archer, 2011; Zhang, Dong, & El Saddik, 2016). A lack of strength in the core or scapular stabilizer muscles during the plank may cause the person to adopt an incorrect posture by compensating with the thoracic spine or lower hips. In fact, a case report indicated that incorrect and excessive scapular activity during plank exercises may lead to long thoracic nerve injury (Güzel, Ozen, & Sözay, 2023). There are studies in the literature examining the activity of the serratus anterior muscle, which is responsible for scapular stabilization, in athletes during plank exercises (Can, Harput, & Turgut, 2024). However, no research has been found that evaluates serratus anterior EMG activity during plank exercises in athletes with scapular dyskinesia."

ELIGIBILITY:
Inclusion Criteria:

* Female athletes aged 13-18 years.

Exclusion Criteria:

* Shoulder pain severe enough to interfere with activity in the past 3 months.
* History of shoulder surgery or fractures.
* Recent acute orthopedic injuries to the lower extremities, upper extremities, or lower back.
* History of any neurological or systemic diseases.
* Significant spinal deformities, such as scoliosis.

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: adolescent athlete
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Surface EMG | baseline
  A NeuroTrac Myoplus Pro (Quintet, Bergen, Norway) EMG device will be used for surface electromyography analysis of the serratus anterior. Disposable 30 x 30 mm round adhesive electrodes will be placed on the dominant side at the 7th intercostal space and at the level of the xiphoid process, while the reference electrode will be positioned on the sternal notch of the sternum. To minimize the negative effects of possible skin movement during the plank exercises, electrodes will be applied while the participant is seated with the trunk in a neutral position and arms flexed at 90 degrees (Januario, Cid, Zanca, Mattiello, & Oliveira, 2022; Konrad, 2005). Participants will perform front plank, prone plank, and side plank exercises for 30 seconds each. Parameters related to muscle strength, total work, and resting tone will be displayed on the device in microvolts, and maximal voluntary contraction will recorded as a percentage.

SECONDARY OUTCOMES:
Core Strength | baseline
  Core endurance in athletes will be assessed using McGill's core endurance tests (McGill, Childs, & Liebenson, 1999). Trunk Flexor Endurance Test, Trunk Extensor Endurance Test and Trunk Lateral Endurance Test will be used for assesment. The time the athlete can maintain this position will be recorded in seconds.
Shoulder rotator strength | baseline
  The internal and external rotation muscle strength of athletes will be assessed using a hand dynamometer with demonstrated reliability (Chamorro, Arancibia, Trigo, Arias-Poblete, & Jerez-Mayorga, 2021). The assessment will be conducted with the athlete in a prone position, with the arm at 90 degrees of abduction and the shoulder in neutral, while the elbow is flexed at 90 degrees (Coinceicao et al., 2018). The dynamometer will be placed proximal to the ulnar styloid process, and the evaluator will stabilize the arm by holding the upper arm with their other hand. The athlete will perform an isometric contraction for 5 seconds. After a 30-second rest, the measurement will be repeated. Each measurement will be conducted three times, and the best score will be recorded. The external rotation/internal rotation (ER/IR) ratio will be calculated using the formula: (External rotation strength / Internal rotation strength) x 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conceicao A, Parraca J, Marinho D, Costa M, Louro H, Silva A, Batalha N. Assessment of isometric strength of the shoulder rotators in swimmers using a handheld dynamometer: a reliability study. Acta Bioeng Biomech. 2018;20(4):113-119. PMID 30821280
- [Background] Cobanoglu, G., Suner Keklik, S., Zorlular, A., Aygun Polat, E., &amp; Akaras, E. (2021). The relationship between scapular and core muscle endurance in professional athletes . Annals of Medical Research, 26(7), 1295-1300. Retrieved from https://annalsmedres.org/index.php/aomr/article/view/1278
- [Background] Topçu, Huseyin, Arabacı, Ramiz, Güngör, Ali Kamil, Birinci, Yakup Zühtü, Pancar, Serkan, &amp;amp; Şekir, Ufuk. (2022). Muscle activity of kore muscles during plank exercise on different surfaces. Turkish Journal of Sport and Exercise, 24(3), 298-305.
- [Background] Neporent, Liz, Schlosberg, Suzanne, &amp;amp;amp; Archer, Shirley J. (2011). Weight training for dummies: John Wiley &amp;amp;amp; Sons.
- [Background] Konrad, Peter. (2005). The abc of emg. A practical introduction to kinesiological electromyography, 1(2005), 30-35.
- [Background] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Background] Kibler WB, Sciascia A. Evaluation and Management of Scapular Dyskinesis in Overhead Athletes. Curr Rev Musculoskelet Med. 2019 Dec;12(4):515-526. doi: 10.1007/s12178-019-09591-1. PMID 31760624
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] da Silva LA, Checchia CS, Goncalves GV, Conte LHG, Santana DS, Barela AMF. EVALUATION OF SCAPULAR DYSKINESIS IN CROSSFIT(R)- PRACTICING ATHLETES. Acta Ortop Bras. 2022 Dec 2;30(spe2):e251074. doi: 10.1590/1413-785220223002e251074. eCollection 2022. PMID 36506859
- [Background] Uga D, Nakazawa R, Sakamoto M. Strength and muscle activity of shoulder external rotation of subjects with and without scapular dyskinesis. J Phys Ther Sci. 2016 Apr;28(4):1100-5. doi: 10.1589/jpts.28.1100. Epub 2016 Apr 28. PMID 27190434
- [Background] Tooth C, Gofflot A, Schwartz C, Croisier JL, Beaudart C, Bruyere O, Forthomme B. Risk Factors of Overuse Shoulder Injuries in Overhead Athletes: A Systematic Review. Sports Health. 2020 Sep/Oct;12(5):478-487. doi: 10.1177/1941738120931764. Epub 2020 Aug 6. PMID 32758080
- [Background] Ludewig PM, Cook TM. Translations of the humerus in persons with shoulder impingement symptoms. J Orthop Sports Phys Ther. 2002 Jun;32(6):248-59. doi: 10.2519/jospt.2002.32.6.248. PMID 12061706
- [Background] Kuniki M, Iwamoto Y, Konishi R, Kuwahara D, Yamagiwa D, Kito N. Neural Drive and Motor Unit Characteristics of the Serratus Anterior in Individuals With Scapular Dyskinesis. J Musculoskelet Neuronal Interact. 2024 Jun 1;24(2):148-158. PMID 38825997
- [Background] Kamonseki DH, Haik MN, Ribeiro LP, Almeida RF, Camargo PR. Scapular movement training is not superior to standardized exercises in the treatment of individuals with chronic shoulder pain and scapular dyskinesis: randomized controlled trial. Disabil Rehabil. 2023 Sep;45(18):2925-2935. doi: 10.1080/09638288.2022.2114552. Epub 2022 Aug 24. PMID 36000960
- [Background] Jildeh TR, Ference DA, Abbas MJ, Jiang EX, Okoroha KR. Scapulothoracic Dyskinesis: A Concept Review. Curr Rev Musculoskelet Med. 2021 Jun;14(3):246-254. doi: 10.1007/s12178-021-09705-8. Epub 2021 Apr 6. PMID 33822304
- [Background] Januario LB, Cid MM, Zanca GG, Mattiello SM, Oliveira AB. Serratus anterior sEMG - sensor placement and test position for normalization purposes during maximal and submaximal exertions. Med Eng Phys. 2022 Mar;101:103765. doi: 10.1016/j.medengphy.2022.103765. Epub 2022 Feb 8. PMID 35232545
- [Background] Huang TS, Chen WJ, Du WY, Lin JJ. Measurement of scapular prominence in symptomatic dyskinesis using a novel scapulometer: reliability and the relationship to shoulder dysfunction. J Shoulder Elbow Surg. 2020 Sep;29(9):1852-1858. doi: 10.1016/j.jse.2020.01.069. Epub 2020 Apr 1. PMID 32247722
- [Background] Guzel S, Ozen S, Sozay S. Scapula winging secondary to prone plank exercise: a case report. Int J Neurosci. 2023 Apr;133(4):426-429. doi: 10.1080/00207454.2021.1924710. Epub 2022 Apr 6. PMID 33930995
- [Background] Fredericson M, Moore T. Muscular balance, core stability, and injury prevention for middle- and long-distance runners. Phys Med Rehabil Clin N Am. 2005 Aug;16(3):669-89. doi: 10.1016/j.pmr.2005.03.001. PMID 16005399
- [Background] Costa E Silva Cabral AL, Marques JP, Dionisio VC. Scapular dyskinesis and overhead athletes: A systematic review of electromyography studies. J Bodyw Mov Ther. 2024 Jul;39:606-614. doi: 10.1016/j.jbmt.2024.03.014. Epub 2024 Mar 16. PMID 38876694
- [Background] Cools AM, Struyf F, De Mey K, Maenhout A, Castelein B, Cagnie B. Rehabilitation of scapular dyskinesis: from the office worker to the elite overhead athlete. Br J Sports Med. 2014 Apr;48(8):692-7. doi: 10.1136/bjsports-2013-092148. Epub 2013 May 18. PMID 23687006
- [Background] Cools AM, Johansson FR, Borms D, Maenhout A. Prevention of shoulder injuries in overhead athletes: a science-based approach. Braz J Phys Ther. 2015 Sep-Oct;19(5):331-9. doi: 10.1590/bjpt-rbf.2014.0109. Epub 2015 Sep 1. PMID 26537804
- [Background] Chamorro C, Arancibia M, Trigo B, Arias-Poblete L, Jerez-Mayorga D. Absolute Reliability and Concurrent Validity of Hand-Held Dynamometry in Shoulder Rotator Strength Assessment: Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Sep 3;18(17):9293. doi: 10.3390/ijerph18179293. PMID 34501883
- [Background] Can EN, Harput G, Turgut E. Shoulder and Scapular Muscle Activity During Low and High Plank Variations With Different Body-Weight-Bearing Statuses. J Strength Cond Res. 2024 Feb 1;38(2):245-252. doi: 10.1519/JSC.0000000000004622. Epub 2023 Oct 8. PMID 37815235
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944